CLINICAL TRIAL: NCT00711100
Title: Preference, Health Effects and Efficacy of Four Oral Tobacco Products for Smoking Cessation
Brief Title: Evaluation of Oral Tobacco as a Harm Reduction Method for Smokers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Minnesota (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 0712M22343; 1R01CA135884 (NIH)
Record Dates: First submitted 2008-07-02; First posted 2008-07-08 (Estimated); Results first posted 2015-09-16 (Estimated); Last update posted 2019-11-18 (Actual); Status verified 2019-10

CONDITIONS: Tobacco Use Disorder
Keywords: Substitution for cigarettes; Oral tobacco products
MeSH Terms: conditions — Tobacco Use Disorder | interventions — stwl protein, Drosophila

STUDY DESIGN:
Masking Description: Open label trial
Oversight: Data Monitoring Committee: Yes

ARMS (5):
- Camel Snus (Experimental): Camel Snus (oral smokeless tobacco product). Dosage: 1.74-1.97 mg nicotine per portion.
  Interventions: Other: Camel Snus
- Marlboro Snus (Experimental): Marlboro Snus (oral smokeless tobacco product). Dosage: 0.14 - 0.38 mg nicotine per portion.
  Interventions: Other: Marlboro Snus
- Stonewall (Experimental): Stonewall (oral dissolvable tobacco product). Dosage: 0.28-0.57 mg nicotine per portion.
  Interventions: Other: Stonewall
- Ariva (Experimental): Ariva (oral dissolvable tobacco product). Dosage: 0.24-0.25 mg nicotine per portion.
  Interventions: Other: Ariva
- General Snus (Experimental): General Snus (oral smokeless tobacco product); Dosage: 3.37 mg nicotine.
  Interventions: Other: General Snus

INTERVENTIONS:
Other: Camel Snus — All subjects will sample Camel Snus and determine if they would prefer to use this product during the abstinence phase over the other products sampled. Sampling period (duration: 1/2 day) requires use of at least 3 samples of Camel Snus. Intervention period (duration: 2 weeks) involves ad libitum daily use (if Camel Snus is chosen for use) during abstinence phase.
  Arms: Camel Snus
Other: Marlboro Snus — All subjects will sample Marlboro Snus and determine if they would prefer to use this product during the abstinence phase over the other products sampled. Sampling period (duration: 1/2 day) requires use of at least 3 samples of Marlboro Snus. Intervention period (duration: 2 weeks) involves ad libitum daily use (if Marlboro Snus is chosen for use) during abstinence phase.
  Arms: Marlboro Snus
Other: Stonewall — All subjects will sample Stonewall and determine if they would prefer to use this product during the abstinence phase over the other products sampled. Sampling period (duration: 1/2 day) requires use of at least 3 samples of Stonewall. Intervention period (duration: 2 weeks) involves ad libitum daily use (if Stonewall is chosen for use) during abstinence phase.
  Arms: Stonewall
Other: Ariva — All subjects will sample Ariva and determine if they would prefer to use this product during the abstinence phase over the other products sampled. Sampling period (duration: 1/2 day) requires use of at least 3 samples of Ariva. Intervention period (duration: 2 weeks) involves ad libitum daily use (if Ariva is chosen for use) during abstinence phase.
  Arms: Ariva
Other: General Snus — All subjects will sample General Snus and determine if they would prefer to use this product during the abstinence phase over the other products sampled. Sampling period (duration: 1/2 day) requires use of at least 3 samples of General Snus. Intervention period (duration: 2 weeks) involves ad libitum daily use (if General Snus is chosen for use) during abstinence phase.
  Arms: General Snus

SUMMARY:
Recently, tobacco companies have developed new oral tobacco products that are purportedly less harmful than conventional tobacco products. These products have not been tested by independent research for their health effects or consumer palatability. In addition, it is not known if these products will be used in addition to cigarette smoking or as a substitute to cigarettes. These two studies will examine four oral tobacco products to answer some of these questions.

The goals of this first study will be to examine: 1) the brand of oral tobacco products which is preferred by cigarette smokers and the pattern and amount of product use when used as a switching tool; 2) the characteristics that are associated with product choice; 3) nicotine exposure from these products; and 4) the withdrawal symptoms from the tobacco products and potential for continued use.

Specifically, our primary aims hypotheses were: 1) the product that will be chosen by most smokers will be based on taste and sensory aspects of the product with products higher in nicotine content more likely to be chosen as the preferred product; and 2) subjects will experience no difficulty using the product for complete cigarette substitution, but a small minority will engage in dual product use.

For the secondary aims, we hypothesized: 1) that compared to the subjects' own brand of cigarettes, the biomarkers for exposure for the oral tobacco products will be significantly lower; 2) withdrawal symptoms from the oral products are likely to occur, but are likely to be mild compared to cigarette withdrawal.

DETAILED DESCRIPTION:
This study will be accomplished by allowing subjects to sample the products and choose one oral tobacco product that they will use instead of cigarettes for a two week period. After the two weeks, they will discontinue all tobacco use and withdrawal symptoms and abstinence rates will be observed.

Subjects will attend an orientation visit where the study will be explained in detail. Interested subjects will sign a consent form and be scheduled to return for baseline measures. Subjects will have a review of medical history to verify that they are in generally good health and do not have contraindications to the study products. Eligible subjects will collect one week of baseline measures while smoking at their normal rate: measures include daily diaries of smoking, questionnaires and urine samples. At the second baseline visit, they will receive samples of the oral tobacco products. The tobacco products tested are five novel oral products recently introduced to the market: 1) Camel Snus (higher nicotine); 2) General Snus (higher nicotine); 3) Marlboro Snus (lower nicotine); and two compressed tobacco tablets, 4) Ariva (lower nicotine), or 5) Stonewall (higher nicotine). All of these tobacco products are purported to have reduced levels of tobacco-specific nitrosamines.

During sample weeks, subjects will be given 10 pouches/tablets of each product in a within-subject design and instructed to use at least three of the daily products in the morning of sample day and resume smoking in the afternoon and through the following day. They will sample the next product in a similar manner. The order of product was randomized. All subjects will sample all five products. This design will allow a short, but adequate trial of each product to determine preference. After the sampling weeks, subjects will choose the product they will want to use to quit smoking. They will be supplied that product over the next two weeks.

During the two weeks of product use during smoking abstinence, subjects will come to weekly clinic visits and then a follow-up visits at 1 week and a phone call at 4 weeks after the end of treatment. At baseline, and 2 weeks post cigarette cessation, subjects will bring in a urine sample from their first morning void and bloods will be drawn. At each visit, subjects will have vital signs obtained (blood pressure, heart rate, weight and carbon monoxide level), they will complete several subjective forms regarding tobacco use, withdrawal symptoms, and mood. Subjects will receive brief behavioral counseling for smoking cessation at all visits.

In addition, during the sample weeks and at the end of two weeks of study product use, subjects will submit three used chews that will be sent to CDC to be analyzed for the tobacco constituents.

ELIGIBILITY:
Inclusion Criteria:

* Cigarette smokers who smoke 10 or more cigarettes per day
* Generally good health

Exclusion Criteria:

* Unstable medical or psychiatric condition.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 104 (Actual)
Dates: Start 2008-08; Primary Completion 2009-10 (Actual); Study Completion 2010-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Dorothy Hatsukami, Ph.D., Principal Investigator — University of Minnesota
Locations (2):
- United States (2):
  - Univeristy of Minnesota, Minneapolis, Minnesota
  - Oregon Research Institute, Eugene, Oregon

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were recruited 10/2008 through 8/2009 through local advertisements in Minnesota and Oregon.
Pre-assignment Details: Sampling Phase preceded the 2 week Abstinence Phase. Sampling phase involved sampling each study product for a 1/2 day; subjects then chose the product that they would like to use for a two week cigarette abstinence period
Groups:
- Oral Tobacco Products: Camel Snus, Marlboro Snus, General Snus, Stonewall, Ariva
Period: Overall Study
Arm/Group | Oral Tobacco Products
Started | 104
Completed | 91
Not Completed | 13
Not completed — Lack of Efficacy | 5
Not completed — Withdrawal by Subject | 8

BASELINE CHARACTERISTICS:
Arm/Group | Oral Tobacco Products
Number analyzed (Participants) | 104
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 2
  Between 18 and 65 years | 97
  >=65 years | 5
Age, Continuous [Mean (Standard Deviation); unit: years] | 40.1 (13.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 40
  Male | 64
Region of Enrollment [Number; unit: participants]
  United States | 104

OUTCOME MEASURES:

1. Primary Outcome: Product Preference
Description: Number of individuals who selected each of the products (e.g., Camel Snus, Marlboro Snus, General Snus, Ariva, Stonewall).
Time Frame: 2 weeks
Measure: Number; unit: participants
Groups:
- Camel Snus: Number of participants who sampled Camel Snus
- Marlboro Snus: Number of participants who sampled Marlboro Snus
- Stonewall: Number of participants who sampled Stonewall
- Ariva: Number of participants who sampled Ariva
- General Snus: Number of partiicipants who sampled General Snus
Arm/Group | Camel Snus | Marlboro Snus | Stonewall | Ariva | General Snus
Number analyzed (Participants) | 98 | 98 | 98 | 98 | 98
participants | 27 | 23 | 24 | 24 | 0

2. Primary Outcome: Abstinence From Cigarettes
Description: Abstinence from cigarettes during Abstinence Phase.
Time Frame: Survival (abstinence) at 3 weeks (2 weeks intervention and 1 week follow-up)
Population: At the end of Sampling Phase, subjects chose a preferred product to use during a two week Abstinence Phase. Abstinence from cigarettes was determined during the 2 week study product phase (e.g., Abstinence Phase) and 1 week after this phase.
Measure: Count of Participants; unit: Participants
Groups:
- Camel Snus; Marlboro Snus; Stonewall; Ariva: Number of participants who preferred this product during abstinence phase
Arm/Group | Camel Snus | Marlboro Snus | Stonewall | Ariva
Number analyzed (Participants) | 27 | 23 | 24 | 24
Participants | 12 | 8 | 5 | 3

ADVERSE EVENTS:
Time Frame: 3 weeks
Groups:
- Camel Snus: Participant who sampled Camel Snus
- Marlboro Snus: Participants who sampled Marlboro Snus
- Stonewall: Participants who sampled Stonewall
- Ariva: Participants who sampled Ariva
- General Snus: Participants who sampled General Snus
Arm/Group | Camel Snus | Marlboro Snus | Stonewall | Ariva | General Snus
Serious Adverse Events (participants affected / at risk) | 0/98 | 0/98 | 0/98 | 0/98 | 0/98
Other Adverse Events (participants affected / at risk) | 9/98 | 5/98 | 9/98 | 5/98 | 23/98
OTHER ADVERSE EVENTS (reported when occurring in more than 3% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Camel Snus (N=98) | Marlboro Snus (N=98) | Stonewall (N=98) | Ariva (N=98) | General Snus (N=98)
Dry Mouth (General disorders) | 1 (1) | 2 (2) | 3 (3) | 1 (1) | 0 (0)
Excessive Salivation (General disorders) | 6 (6) | 2 (2) | 1 (1) | 2 (2) | 14 (14)
Dizziness/Lightheadedness (General disorders) | 0 (0) | 0 (0) | 3 (3) | 1 (1) | 3 (3)
Sore Throat (General disorders) | 2 (2) | 1 (1) | 2 (2) | 1 (1) | 6 (6)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No